CLINICAL TRIAL: NCT02785055
Title: Evaluation of Ultrasound-Assisted Thoracic Epidural Placement in Patients Undergoing Upper Abdominal and Thoracic Surgery: A Randomized, Double-Blind Study
Brief Title: Neuraxial Ultrasound for Thoracic Epidural Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benaroya Research Institute (Other)
Responsible Party: Principal Investigator, David Auyong, Anesthesiologist, Benaroya Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB08130
Record Dates: First submitted 2016-05-18; First posted 2016-05-27 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Analgesia, Epidural
MeSH Terms: conditions — Agnosia | interventions — Hydromorphone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound-Assisted (Active Comparator): Ultrasound assisted marking of the thoracic spine on the skin for Thoracic Epidural Placement
  Interventions: Procedure: Thoracic Epidural Placement; Drug: Bupivacaine 0.05%; Drug: Hydromorphone 0.01mg/mL
- Palpation (Active Comparator): Palpation marking of the thoracic spine on the skin for Thoracic Epidural Placement
  Interventions: Procedure: Thoracic Epidural Placement; Drug: Bupivacaine 0.05%; Drug: Hydromorphone 0.01mg/mL

INTERVENTIONS:
Procedure: Thoracic Epidural Placement — Thoracic Epidural Placement
Drug: Bupivacaine 0.05% — Delivery of epidural solution containing both bupivacaine 0.05%/hydromorphone0.01mg/mL solution
Drug: Hydromorphone 0.01mg/mL — Delivery of epidural solution containing both bupivacaine 0.05%/hydromorphone0.01mg/mL solution

SUMMARY:
This blinded, randomized study compares standard palpation to ultrasound-assisted landmark identification of the thoracic spine for thoracic epidural catheterization.

DETAILED DESCRIPTION:
In this study, the investigators will utilize ultrasonography to identify midline bony landmarks including spinous processes, laminae, and intervertebral interspaces prior to the initial needle placement and compare this to standard palpation of the bony thoracic spine for thoracic epidural placement. The investigators will evaluate and compare the two needle localization techniques by the following outcomes: time to identify the epidural space by loss of resistance, needle passes, skin punctures, recovery room pain scores, and epidural success.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology Classification I-IV
* thoracic surgery
* abdominal surgery

Exclusion Criteria:

* contraindications to epidural catheter
* pregnancy
* coagulopathy
* infection (localized)
* allergy to local anesthetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-04; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Time to epidural space identification | Estimated 10 minutes
  Needle insertion through the skin until loss-of-resistance with slip syringe, evaluated by a blinded individual reviewing a video recording of the procedure.

SECONDARY OUTCOMES:
Needle passes | Estimated 10 minutes
  Attempt to place needle into the interlaminar foramina. Needle tip movements toward midline and cephalad were counted as s single pass. Additional passes were counted when the needle was returned to a plane parallel to the skin.
Needle skin punctures | Estimated 10 minutes
  Complete needle withdrawal from the skin and re-insertion at new location
Pain Score | Through study completion, estimated 4 hours
  Numeric rating scale pain score on recovery room arrival, prior to IV analgesics.
Working epidural | Through study completion, estimated 4 hours
  Loss of temperature discrimination to ice and pain score <= 5.

CONTACTS AND LOCATIONS:
Overall Officials: David Auyong, MD, Principal Investigator — Virginia Mason Medical Center
Locations (1):
- Virginia Mason Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided
No Plan in place

REFERENCES:
- [Derived] Auyong DB, Hostetter L, Yuan SC, Slee AE, Hanson NA. Evaluation of Ultrasound-Assisted Thoracic Epidural Placement in Patients Undergoing Upper Abdominal and Thoracic Surgery: A Randomized, Double-Blind Study. Reg Anesth Pain Med. 2017 Mar/Apr;42(2):204-209. doi: 10.1097/AAP.0000000000000540. PMID 28002229